CLINICAL TRIAL: NCT01929681
Title: Low Field Magnetic Stimulation in Mood Disorders: Three Daily Visits
Brief Title: Multiple Treatment Study Using Low Field Magnetic Stimulation for Bipolar Depression
Acronym: LFMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other)
Responsible Party: Principal Investigator, Michael Rohan, Imaging Physicist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012P002380
Record Dates: First submitted 2013-07-23; First posted 2013-08-28 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Bipolar Depression
Keywords: Low Field Magnetic Stimulation; bipolar; depression; alternative treatment
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LFMS - active treatment (Experimental): Low Field Magnetic Stimulation (LFMS) active treatment
  Active low field magnetic stimulation treatment applied with the LFMS Device; the device is on and magnetic field stimulation is present.
  Interventions: Device: Low Field Magnetic Stimulation
- LFMS - sham treatment (Sham Comparator): Low Field Magnetic Stimulation - sham treatment
  Inactive low field magnetic stimulation (no stimulation) treatment applied with the LFMS Device; the device is on, however no magnetic field stimulation is present.
  Interventions: Device: Low Field Magnetic Stimulation

INTERVENTIONS:
Device: Low Field Magnetic Stimulation — Low Field Magnetic Stimulation is an electromagnetic technique. It uses low strength electric fields operating at a high frequency.
  Other Names: LFMS

SUMMARY:
Objectives:

To demonstrate the duration of the antidepressant effect of Low Field Magnetic Stimulation (LFMS)in subjects with bipolar depression.

Hypotheses:

Investigators expect subjects who receive LFMS to show significant mood improvement one week after the start of a three day course of daily stimulation as compared to subjects who receive sham LFMS.

Investigators expect subjects who receive LFMS to show immediate mood improvement over the first treatment as measured by the difference in pre and post-treatment PANAS+ ratings.

Investigators expect to show that LFMS will be well tolerated in a three-treatment protocol.

DETAILED DESCRIPTION:
Low Field Magnetic Stimulation is an electromagnetic intervention being investigated at McLean Hospital because of its effect on symptoms of depression. It consists of pulsed electric fields that are induced remotely in the head by a portable coil. It has been observed to have mood elevating effects in depressed patients with Bipolar Disorder (BPD). These effects are immediate, occurring upon completion of a 20 minute treatment.

LFMS is unique because of its low electric field strength, and because of its high frequency operation, compared to other electromagnetic treatments. While other treatments such as Electroconvulsive Therapy (ECT) use electric fields equivalent to > 100-200 Volts/meter to affect the brain, LFMS uses <1 V/m. Such a low electric field strength indicates that another mechanism is activated by LFMS, and this provides a possibility for a new treatment. It may also give insight into causes of depression.

LFMS is also unique because it has an immediate effect. This immediate effect may have implications for emergency treatment.

The purpose of this study is to observe the response to LFMS in depressed BPD subjects with the aim of assessing the effects of multiple treatments, and of observing the duration of the mood improvement.To do so, the investigators propose to study 72 subjects in a protocol of three treatments in three days. Subjects will be rated before and after each treatment, and will return for mood ratings at one week after treatment. Investigators hope that this characterization of LFMS will allow clinical research groups to perform large trials and to evaluate its clinical effectiveness in patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be men or women between the ages of 21-65.
2. Subjects must not have serious physical illnesses, neurological diseases or dementias.
3. Subjects will meet DSM-IV criteria for Bipolar Disorder Type I or II and meet criteria for current depression (DSM-IV major depressive episode, current).
4. Subject must have a MADRS >= 20, Young Mania Rating Score (YMRS score) < 7.
5. Subjects must be capable of providing informed consent.
6. Subjects must have an established residence and phone.
7. Subjects may be medicated or unmedicated.

Exclusion Criteria:

1. Dangerous or active suicidal ideation.
2. Pregnant or planning on becoming pregnant.
3. Substance abuse (cannot meet DSM criteria for substance abuse, no significant drug abuse within last 3 months, no major polysubstance abuse history, no history of dependence in last year, no drug use within last month).
4. Mania, hypomania or mixed mood state.
5. Significant medical or neurological illness that might pose a risk to study enrollment or interfere with interpretation of study data.
6. Changes in psychiatric medication (e.g. dose or drug) within 6 weeks prior to enrollment.
7. History of schizophrenia, schizoaffective, obsessive-compulsive or post-traumatic stress disorders.
8. Treatment resistant depression (as determined by the study psychiatrist; consistently and substantially symptomatic over several years despite electroconvulsive therapy, 2 or more adequate trials of a primary mood stabilizer with antidepressant effects (e.g., lithium, valproate or lamotrigine) or antidepressant medications (e.g., bupropion, Selective Serotonin Reuptake Inhibitors (SSRI) or Serotonin Norepinephrine Reuptake Inhibitor (SNRI).)
9. Contraindications for Magnetic Resonance Imaging (MRI): Presence of a pacemaker, neurostimulator, or metal in head or neck.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Rohan, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed through newspaper advertisement, posting, and referral
Pre-assignment Details: Subjects that failed exclusion criteria for variable criteria such as medications change or drug use were permitted to reapply for participation after a washout period of at least 1 month.
Groups:
- LFMS - Active Treatment: Low Field Magnetic Stimulation (LFMS) active treatment
  Active low field magnetic stimulation treatment applied with the LFMS Device; the device is on and magnetic field stimulation is present.
  Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic technique. It uses low strength electric fields operating at a high frequency.
- LFMS - Sham Treatment: Low Field Magnetic Stimulation - sham treatment
  Inactive low field magnetic stimulation (no stimulation) treatment applied with the LFMS Device; the device is on, however no magnetic field stimulation is present.
  Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic technique. It uses low strength electric fields operating at a high frequency.
Period: Overall Study
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment
Started | 28 | 25
Completed | 26 | 24
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Three enrolled subjects did not complete.
Groups:
- Total: Total of all reporting groups
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.5) | 45.7 (10.3) | 45.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 15 | 15 | 30
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating scale assesses 10 symptom areas of depression during an interview. Each of the 10 items received a score ranging from 0 to 6. The scale has a range of 0-60 for the reported total.
  units on a scale | 28.2 (5.8) | 27.4 (5.0) | 27.8 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Long Term Change: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: The Montgomery-Asberg Depression Rating scale assesses 10 symptom areas of depression during an interview. Each of the 10 items received a score ranging from 0 to 6. The scale has a range of 0-60 for the reported total. A higher score indicates increased depression for all items and for the total. This outcome measure is the change from pretreatment baseline acquired at the screening visit to a follow-up visit 7 days after the first treatment.
Time Frame: Variable based on screening visit schedule, > 2 weeks.
Population: Subjects completing 3 treatments and 1 visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment
Number analyzed (Participants) | 26 | 24
units on a scale | -14.03 (7.85) | -9.75 (9.32)
Statistical Analysis 1: Comparison: LFMS - Active Treatment vs LFMS - Sham Treatment; Test type: Superiority; p < 0.049, Regression, Linear

2. Primary Outcome: Change Over First Treatment: Positive and Negative Affect Schedule (PANAS) Positive Items Subscale
Description: PANAS consists of 10 positive and 10 negative valence word items. Items are rated by the participant to indicate their assessment of how they are feeling about this item "right now" on a scale of 1(slightly) or not at all through 5 (extremely). 10 of of the items form a positive affect subscale, in which a higher score indicates increased positive affect, with a subscale range of 10 to 50. 10 of the items form a negative affect subscale, in which a higher score indicates more negative affect, with a subscale range of 10 to 50. This outcome measure is change in the 10 item positive affect subscale. This outcome measure is the difference between the scale administered immediately (<30min) prior to the first treatment and immediately after (<30min) the first treatment.
Time Frame: 90 minutes; change immediately (<30min) prior to the first treatment and immediately after (<30min) the first treatment.
Population: subjects completing 3 treatment visits and 1 followup visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment
Number analyzed (Participants) | 26 | 24
units on a scale | 0.5 (5.8) | 1.4 (5.32)
Statistical Analysis 1: Comparison: LFMS - Active Treatment vs LFMS - Sham Treatment; Test type: Superiority; p < 0.182, Regression, Linear

3. Secondary Outcome: Rate of of Change in Daily Improvement Over 3 Treatments: Positive and Negative Affect Schedule (PANAS) Positive Items Subscale
Description: PANAS consists of 10 positive and 10 negative valence word items. Items are rated by the participant to indicate their assessment of how they are feeling about this item "right now" on a scale of 1(slightly) or not at all through 5 (extremely). 10 of of the items form a positive affect subscale, in which a higher score indicates increased positive affect, with a subscale range of 10 to 50. 10 of the items form a negative affect subscale, in which a higher score indicates more negative affect, with a subscale range of 10 to 50. This outcome measure uses the 10 item positive affect subscale. This outcome measure is the least squares fit of a linear coefficient to the three post (<30min oost treatment) minus pre (<30min pre treatment) score differences for the three treatment days
Time Frame: Over 3 days of treatment
Population: Subjects completing 3 treatments and 1 visit
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment
Number analyzed (Participants) | 26 | 24
units on a scale
  linear coefficient | -0.471 (0.594) | -0.375 (0.648)
  day 1 mean | 0.50 (1.14) | 1.40 (1.09)
  day 2 mean | -0.63 (0.68) | 0.21 (0.91)
  day 3 mean | -0.44 (0.65) | 0.65 (0.77)
Statistical Analysis 1: Comparison: LFMS - Active Treatment vs LFMS - Sham Treatment; Test type: Superiority; p < 0.449, Regression, Linear; Mixed effects analysis

4. Secondary Outcome: Rate of Change Over 3 Treatments: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Asberg Depression Rating scale assesses 10 symptom areas of depression during an interview. Each of the 10 items received a score ranging from 0 to 6. The scale has a range of 0-60 for the reported total. A higher score indicates increased depression for all items and for the total. This outcome measure is the least squares fit of a linear coefficient to the three pretreatment scores for the three treatment days
Time Frame: Over 3 days of treatment
Population: Subjects completing 3 treatments and 1 visit
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment
Number analyzed (Participants) | 26 | 24
units on a scale
  linear coefficient | -5.42 (1.07) | -5.60 (1.07)
  day 1 mean | 26.15 (1.47) | 26.13 (1.44)
  day 2 mean | 16.81 (1.31) | 17.83 (1.45)
  day 3 mean | 15.31 (1.69) | 14.92 (1.66)
Statistical Analysis 1: Comparison: LFMS - Active Treatment vs LFMS - Sham Treatment; Test type: Superiority; p < 0.444, Regression, Linear; Mixed effects analysis

5. Secondary Outcome: Rate of Change Over 3 Treatments: Positive and Negative Affect Schedule (PANAS) Positive Items Subscale
Description: PANAS consists of 10 positive and 10 negative valence word items. Items are rated by the participant to indicate their assessment of how they are feeling about this item "right now" on a scale of 1(slightly) or not at all through 5 (extremely). 10 of of the items form a positive affect subscale, in which a higher score indicates increased positive affect, with a subscale range of 10 to 50. 10 of the items form a negative affect subscale, in which a higher score indicates more negative affect, with a subscale range of 10 to 50. This outcome measure uses the 10 item positive affect subscale. This outcome measure is the least squares fit of a linear coefficient to the three pretreatment scores for the three treatment days
Time Frame: Over 3 days of treatment
Population: Subjects completing 3 treatments and 1 visit
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment
Number analyzed (Participants) | 26 | 24
units on a scale
  linear coefficient | 1.70 (1.39) | 0.80 (1.10)
  day 1 mean | 21.00 (1.82) | 22.25 (1.34)
  day 2 mean | 24.04 (1.95) | 23.54 (1.53)
  day 3 mean | 24.40 (2.21) | 23.85 (1.84)
Statistical Analysis 1: Comparison: LFMS - Active Treatment vs LFMS - Sham Treatment; Test type: Superiority; p < 0.182, Regression, Linear; Mixed effects analysis

ADVERSE EVENTS:
Time Frame: Adverse events data was collected over a period of 3 years.
Arm/Group | LFMS - Active Treatment | LFMS - Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 1/26 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LFMS - Active Treatment (N=26) | LFMS - Sham Treatment (N=24)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0) — A night of insomnia reported the night after the second of three treatments

LIMITATIONS AND CAVEATS:
Study was designed for 72 subjects but only 50 subjects were completed due to lack of funds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No